CLINICAL TRIAL: NCT07263906
Title: Dose Escalation and Expansion Clinical Study of Targeted LILRA6 CAR-T for the Treatment of Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Clinical Study of LILRA6 CAR-T for the Treatment of R/R Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1003
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-10

CONDITIONS: Refractory Acute Myeloid Leukemia; Recurrent Acute Myeloid Leukemia
Keywords: Refractory/recurrent acute myeloid leukemia; LILRA6 CAR-T; Acute myeloid leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PB LILRA6 CAR-T (Experimental)
  Interventions: Biological: Anti-LILRA6 CAR-T cells

INTERVENTIONS:
Biological: Anti-LILRA6 CAR-T cells — lentiviral vector-transducted peripheral blood-derived T cells to express anti-LILRA6 CAR

SUMMARY:
This study aims to evaluate the safety and efficacy of LILRA6-directed chimeric antigen receptor T cells (LILRA6 CAR-T cells) in patients with refractory or relapsed acute myeloid leukemia(AML).

DETAILED DESCRIPTION:
This is a single-center, open-label, single-arm, dose-escalation and dose-expansion phase I clinical trial designed to evaluate the safety and preliminary efficacy of LILRA6-targeted CAR-T cell therapy in patients with relapsed or refractory acute myeloid leukemia (AML) expressing LILRA6.

Phase I (Dose Escalation) The dose-escalation phase will follow a conventional 3+3 design, with a single dose level administered via intravenous infusion. Each cohort will include 3 to 6 patients. Following the initial infusion, patients will be monitored for at least 28 days to assess safety, and subsequently followed for up to 2 years to evaluate long-term outcomes.

Phase II (Dose Expansion) Based on the safety profile, persistence of LILRA6 CAR-T cells, and preliminary efficacy results observed in Phase I, the recommended dose and administration schedule will be established. Approximately 30 eligible patients will then be enrolled in the dose-expansion phase to further assess the safety and efficacy of LILRA6 CAR-T cell therapy at the selected dose. After the first infusion, all patients will continue in long-term follow-up for up to 2 years post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in this study and sign the informed consent form.
2. Age range: 18 - 75 years old. Gender is not restricted.
3. Refractory/Recurrent AML: Meeting any one of the following criteria for refractory or recurrent cases is sufficient. 1) Refractory: (1) In the case of a newly diagnosed patient, treatment with the standard regimen for two courses fails to achieve complete remission (CR); (2) Recurrence within 12 months after consolidation and intensification therapy following CR; (3) Recurrence after 12 months with no response to salvage chemotherapy; (4) ≥ 2 recurrences; (5) Persistent extramedullary leukemia; 2) Recurrence: (1) Leukemia cells reappear in the peripheral blood after complete remission (CR) of AML; (2) The percentage of blasts in the bone marrow is ≥ 5% (excluding other reasons such as bone marrow regeneration after consolidation chemotherapy); (3) Infiltration of leukemia cells in sites other than the bone marrow (excluding the central nervous system).
4. Expected survival period ≥ 12 weeks.
5. The positive rate of LILRA6 expression in bone marrow/tumor cells is ≥ 20%
6. ECOG score ranging from 0 to 2 points.
7. Sufficient organ function reserve: Alanine aminotransferase and Aspartate aminotransferase ≤ 2.5× UNL (upper limit of normal value); Creatinine clearance rate (Cockcroft-Gault method) ≥ 45 mL/min; Serum total bilirubin ≤ 1.5× UNL; Ejection fraction of the heart (EF) ≥ 45%; In an indoor natural air environment, baseline oxygen saturation > 92%; Blood routine: All of the following criteria are met: Absolute number of neutrophils ≥ 0.5×10^9 /L, Platelet count ≥ 30×10^9 /L, Hemoglobin ≥ 7.0 g/dl.
8. Allow those who have previously undergone a single autologous hematopoietic stem cell transplantationAllowing previous recipients of a single autologous hematopoietic stem cell transplantation.
9. Pregnancy tests for the female subjects of childbearing age must be negative, and they must also agree to take effective contraceptive measures during the trial.
10. There are no uncontrollable infectious activities (including lung infections).
11. Distance from the last anti-tumor treatment: Systemic chemotherapy / systemic radiotherapy / immunotherapy ≥ 3 weeks, targeted drug elution period ≥ 2 weeks.
12. No active infection of the novel coronavirus or influenza.

Exclusion Criteria:

1. Those who have a severe history of allergic reaction to any component of the cell preparation or the pre-treatment chemotherapy drugs.
2. Those with a history of other active malignant tumors.
3. There are active infections that require treatment (excluding simple urinary tract infections and bacterial pharyngitis); the use of prophylactic antibiotics, antiviral drugs, and antifungal drugs is permitted.
4. Active hepatitis B (with HBsAg positive and HBV-DNA ≥ 10³ copies/mL), hepatitis C infection, syphilis, or other acquired/innate immune deficiency disorders (including HIV infection).
5. According to the New York Heart Association (NYHA) classification of cardiac function, those with cardiac function at grade III or IV.
6. Previous anti-tumor treatment-related toxic reactions have not yet recovered to a grade ≤ 1 (according to CTCAE 5.0), except for fatigue, anorexia and hair loss.
7. Those with a history of epilepsy or other central nervous system diseases that may affect the research assessment.

8: Those who have received any other targeted LILRA6 drug treatment before. 9.Breastfeeding women who do not wish to stop breastfeeding. 10.The researchers believe that there may be any other circumstances that could increase the risks for the subjects or interfere with the test results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLTs) | Up to 28 days
  To evaluate the safety, tolerability, and determine the recommended dosage of peripheral blood-derived Anti-LILRA6 CAR-T Cell Therapy for refractory/relapsed peripheral T-cell lymphoma.

SECONDARY OUTCOMES:
Complete response rate (CR) | 3 months
  To determine the anti-tumor effectivity of PB LILRA6 CAR-T

OTHER OUTCOMES:
Overall response rate (ORR) | 3 months
  To determine the anti-tumor effectivity of PB LILRA6 CAR-T
Progression free survival (PFS) | Up to 2 years
  To determine the anti-tumor effectivity of PB LILRA6 CAR-T
Overall survival (OS) | Up to 2 years
  To determine the anti-tumor effectivity of PB LILRA6 CAR-T
Duration of response (DOR) | Up to 2 years
  To determine the anti-tumor effectivity of PB LILRA6 CAR-T

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Qian, Professor, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital,School of Medicine,Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No